CLINICAL TRIAL: NCT03316885
Title: Post-Market Clinical Investigation of the Clareon® IOL
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Alcon Research (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ILJ466-P003
Record Dates: First submitted 2017-10-18; First posted 2017-10-20 (Actual); Results first posted 2023-08-21 (Actual); Last update posted 2023-08-21 (Actual); Status verified 2023-08

CONDITIONS: Cataract; Aphakia
MeSH Terms: conditions — Cataract; Aphakia | interventions — Cataract Extraction

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Clareon IOL (Experimental): Clareon® aspheric hydrophobic acrylic intraocular lens implanted with the Alcon Monarch III-D delivery system as a replacement of the human crystalline lens during cataract surgery
  Interventions: Device: Clareon® IOL; Procedure: Cataract Surgery

INTERVENTIONS:
Device: Clareon® IOL — Foldable, single-piece posterior chamber IOL intended for long-term use over the lifetime of the cataract patient. This device is CE-marked (European Conformity) in the countries with participating Investigators.
  Other Names: Model SY60WF
Procedure: Cataract Surgery — Routine small incision cataract surgery with unilateral IOL implantation

SUMMARY:
The primary purpose of this study is to evaluate the long-term (3 years) visual acuity and adverse event outcomes for the Clareon® Intraocular Lens (IOL). A comparison to historical safety and performance endpoint (SPE) rates as reported in the European Standard International Organization for Standardization (EN ISO) 11979-7:2014 will be conducted at one year. The secondary purpose of this study is to evaluate the visual acuity outcomes with the Clareon IOL at Years 2 and 3.

DETAILED DESCRIPTION:
Subjects will attend a total of 12 study visits over a period of approximately 36 months: One preoperative screening visit, two operative visits, and nine post-implantation visits. Both eyes will be implanted, with the second eye implantation to occur 2-21 days after the first. Primary endpoint data will be collected at the Year 1 visit (Day 330-420 post-implantation from second eye surgery).

ELIGIBILITY:
Key Inclusion Criteria:

* Diagnosed with bilateral cataracts
* Planned small incision cataract removal surgery
* Able to comprehend and willing to sign a statement of informed consent and complete all required post-implantation visits

Key Exclusion Criteria:

* Subjects who may reasonably be expected to require ocular surgical treatment or refractive surgical procedures at any time during the study
* Certain eye conditions, as specified in the protocol, including but not limited to glaucoma, diabetic retinopathy, diabetic macular edema, and macular degeneration
* Pregnant or lactating, current or planned during the course of the study

Other protocol-defined inclusion/exclusion criteria may apply.

Min Age: 22 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 245 (Actual)
Dates: Start 2018-03-14 (Actual); Primary Completion 2019-10-18 (Actual); Study Completion 2021-09-23 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Sr. Clinical Trial Lead, CDMA, Surgical, Study Director — Alcon Research, LLC
Locations (19):
- Australia (3):
  - Alcon Investigative Site, Footscray, Victoria
  - Alcon Investigative Site, Mornington, Victoria
  - Alcon Investigative Site, Sydney
- France (3):
  - Alcon Investigative Site, Brest, Cedex
  - Alcon Investigative Site, Lyon
  - Alcon Investigative Site, Paris
- Germany (2):
  - Alcon Investigative Site, Frankfurt
  - Alcon Investigative Site, Heidelberg
- Italy (2):
  - Alcon Investigative Site, Perugia
  - Alcon Investigative Site, Pisa
- Alcon Investigative Site, Amsterdam, Netherlands
- Spain (5):
  - Alcon Investigative Site, Jerez de la Frontera, Cadiz
  - Alcon Investigative Site, Alcalá de Henares
  - Alcon Investigative Site, Oviedo
  - Alcon Investigative Site, San Sebastián
  - Alcon Investigative Site, Valencia
- United Kingdom (3):
  - Alcon Investigative Site, Sutton, Carshalton
  - Alcon Investigative Site, Brighton
  - Alcon Investigative Site, London

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Study participants were recruited from 19 study centers located in Australia (n = 3), France (n = 2), Germany (n = 2), Italy (n = 2), the Netherlands (n = 2), Spain (n = 5), and the United Kingdom (n = 3).
Pre-assignment Details: Of the 245 enrolled, 30 participants were discontinued from the study prior to attempted implantation with the IOL. This reporting group includes all participants with attempted implantation (215).
Units Other Than Participants: eyes
Period: Overall Study
Arm/Group | Clareon IOL
Started | 215; 430 eyes
Implanted in First Eye Only | 215; 215 eyes
Implanted in Second Eye Only | 209; 209 eyes
Implanted in 1 Eye Only | 6; 6 eyes
Completed | 183; 365 eyes (One participant was monocular at Year 3.)
Not Completed | 32; 65 eyes
Not completed — Adverse Event | 1
Not completed — Death | 10
Not completed — Lost to Follow-up | 4
Not completed — Withdrawal by Subject | 9
Not completed — COVID related | 8

BASELINE CHARACTERISTICS:
Population: All Implanted Analysis Set: All subjects/eyes with successful test article implantation
Arm/Group | Clareon IOL
Number analyzed (Participants) | 215
Age, Continuous [Mean (Standard Deviation); unit: years] | 72.1 (8.07)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 126
  Male | 89
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 17
  Not Hispanic or Latino | 195
  Unknown or Not Reported | 3
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 6
  Native Hawaiian or Other Pacific Islander | 1
  Black or African American | 3
  White | 204
  More than one race | 0
  Other | 1

OUTCOME MEASURES:

1. Primary Outcome: Percentage of First Implanted Eyes Achieving Best-Corrected Distance Visual Acuity (BCDVA) of 0.3 Logarithm Minimum Angle of Resolution (logMAR) or Better at 1 Year Post-Implantation
Description: Visual acuity (VA) was tested for the first implanted eye using the correction obtained from the manifest refraction and 100% contrast electronic Early Treatment Diabetic Retinopathy Study (ETDRS) charts at a distance of 4 meters (m) from the eye. VA was measured in logarithm of the minimum angle of resolution (logMAR), with 0.02 logMAR increment corresponding to a single letter on an ETDRS chart. A BCDVA of 0.3 logMAR is equivalent to 20/40 Snellen visual acuity. VA was compared to the historical safety and performance endpoint (SPE) of 92.5% [as reported in the European Standard International Organization for Standardization (EN ISO) 11979-7:2014].
Time Frame: Year 1 post-implantation from second eye surgery
Population: All Implanted Analysis Set with data
Measure: Number (95% Confidence Interval); unit: percentage of first implanted eyes
Units Other Than Participants: first implanted eye
Arm/Group | Clareon IOL
Number analyzed (Participants) | 198
Number analyzed (first implanted eye) | 198
percentage of first implanted eyes | 99.5 [97.2 to 100.0]
Statistical Analysis 1: Comparison: Clareon IOL; Test type: Other — The performance target in support of the primary effectiveness was percentage of eyes achieving objective monocular BCDVA at 1 year postoperative (Visit 5A) compared to the a priori SPE percentage of 92.5%. This is for the All Implanted Analysis Set (AAS) (as reported in EN ISO 11979-7:2014); Comparison = 100.0, 95% CI 1-sided [upper limit 100.0]

2. Primary Outcome: Percentage of Second Implanted Eyes Achieving BCDVA of 0.3 logMAR or Better at 1 Year Post-Implantation
Description: VA was tested for the second implanted eye using the correction obtained from the manifest refraction and 100% contrast electronic ETDRS charts at a distance of 4 m from the eye. VA was measured in logMAR, with 0.02 logMAR increment corresponding to a single letter on an ETDRS chart. A BCDVA of 0.3 logMAR is equivalent to 20/40 Snellen visual acuity. VA was compared to the historical SPE of 92.5% (EN ISO 11979-7:2014).
Time Frame: Year 1 post-implantation from second eye surgery
Population: All Implanted Analysis Set with data
Measure: Number (95% Confidence Interval); unit: percentage of second implanted eyes
Units Other Than Participants: second implanted eye
Arm/Group | Clareon IOL
Number analyzed (Participants) | 198
Number analyzed (second implanted eye) | 198
percentage of second implanted eyes | 99.5 [97.2 to 100.0]
Statistical Analysis 1: Comparison: Clareon IOL; Test type: Other — [test comment as in outcome 1, analysis 1]; Comparison = 100.0, 95% CI 1-sided [upper limit 100.0]

3. Secondary Outcome: Percentage of First Implanted Eyes Achieving BCDVA of 0.3 logMAR or Better at 2 Years Post-Implantation
Description: VA was tested for the first implanted eye using the correction obtained from the manifest refraction and 100% contrast electronic ETDRS charts at a distance of 4 m from the eye. VA was measured in logMAR, with 0.02 logMAR increment corresponding to a single letter on an ETDRS chart. A BCDVA of 0.3 logMAR is equivalent to 20/40 Snellen visual acuity. No hypothesis testing was prespecified for this endpoint.
Time Frame: Year 2 post-implantation from second eye surgery
Population: All Implanted Analysis Set with data
Measure: Number (95% Confidence Interval); unit: percentage of second implanted eyes
Units Other Than Participants: second implanted eye
Arm/Group | Clareon IOL
Number analyzed (Participants) | 190
Number analyzed (second implanted eye) | 190
percentage of second implanted eyes | 99.5 [97.1 to 100.0]

4. Secondary Outcome: Percentage of Second Implanted Eyes Achieving BCDVA of 0.3 logMAR or Better at 2 Years Post-Implantation
Description: VA was tested for the second implanted eye using the correction obtained from the manifest refraction and 100% contrast electronic ETDRS charts at a distance of 4 m from the eye. VA was measured in logMAR, with 0.02 logMAR increment corresponding to a single letter on an ETDRS chart. A BCDVA of 0.3 logMAR is equivalent to 20/40 Snellen visual acuity. No hypothesis testing was prespecified for this endpoint.
Time Frame: Year 2 post-implantation from second eye surgery
Population: All Implanted Analysis Set with data
Measure: Number (95% Confidence Interval); unit: percentage of second implanted eyes
Units Other Than Participants: second implanted eye
Arm/Group | Clareon IOL
Number analyzed (Participants) | 189
Number analyzed (second implanted eye) | 189
percentage of second implanted eyes | 98.9 [96.2 to 99.9]

5. Secondary Outcome: Percentage of First Implanted Eyes Achieving BCDVA of 0.3 logMAR or Better at 3 Years Post-Implantation
Description: as for outcome 3
Time Frame: Year 3 post-implantation from second eye surgery
Population: All Implanted Analysis Set with data
Measure: Number (95% Confidence Interval); unit: percentage of first implanted eyes
Units Other Than Participants: first implanted eye
Arm/Group | Clareon IOL
Number analyzed (Participants) | 183
Number analyzed (first implanted eye) | 183
percentage of first implanted eyes | 99.5 [97.0 to 100.0]

6. Secondary Outcome: Percentage of Second Implanted Eyes Achieving BCDVA of 0.3 logMAR or Better at 3 Years Post-Implantation
Description: as for outcome 4
Time Frame: Year 3 post-implantation from second eye surgery
Population: All Implanted Analysis Set
Measure: Number (95% Confidence Interval); unit: percentage of second implanted eyes
Units Other Than Participants: second implanted eye
Arm/Group | Clareon IOL
Number analyzed (Participants) | 182
Number analyzed (second implanted eye) | 182
percentage of second implanted eyes | 98.9 [96.1 to 99.9]

7. Secondary Outcome: Uncorrected Distance Visual Acuity (UCDVA) at 1 Year Post-Implantation - First Implanted Eye
Description: VA was tested for the first implanted eye without visual correction using 100% contrast electronic ETDRS charts at a distance of 4 m from the eye. +0.25 diopter (D) spherical power was applied to correct for optical infinity. VA was measured in logMAR, with 0.02 logMAR increment corresponding to a single letter on an ETDRS chart. A UCDVA of 0.0 logMAR is equivalent to 20/20 Snellen visual acuity, with a lower numeric value representing better visual acuity. No hypothesis testing was prespecified for this endpoint.
Time Frame: Year 1 post-implantation from second eye surgery
Population: All Implanted Analysis Set with data
Measure: Mean (Standard Deviation); unit: logMAR
Units Other Than Participants: first implanted eye
Arm/Group | Clareon IOL
Number analyzed (Participants) | 199
Number analyzed (first implanted eye) | 199
logMAR | 0.079 (0.1499)

8. Secondary Outcome: UCDVA at 1 Year Post-Implantation - Second Implanted Eye
Description: VA was tested for the second implanted eye without visual correction using 100% contrast electronic ETDRS charts at a distance of 4 m from the eye. +0.25 D spherical power was applied to correct for optical infinity. VA was measured in logMAR, with 0.02 logMAR increment corresponding to a single letter on an ETDRS chart. A UCDVA of 0.0 logMAR is equivalent to 20/20 Snellen visual acuity, with a lower numeric value representing better visual acuity. No hypothesis testing was prespecified for this endpoint.
Time Frame: Year 1 post-implantation from second eye surgery
Population: All Implanted Analysis Set with data
Measure: Mean (Standard Deviation); unit: logMAR
Units Other Than Participants: second implanted eye
Arm/Group | Clareon IOL
Number analyzed (Participants) | 198
Number analyzed (second implanted eye) | 198
logMAR | 0.058 (0.1364)

9. Secondary Outcome: UCDVA at 2 Years Post-Implantation - First Implanted Eye
Description: VA was tested for the first implanted eye without visual correction using 100% contrast electronic ETDRS charts at a distance of 4 m from the eye. +0.25 D spherical power was applied to correct for optical infinity. VA was measured in logMAR, with 0.02 logMAR increment corresponding to a single letter on an ETDRS chart. A UCDVA of 0.0 logMAR is equivalent to 20/20 Snellen visual acuity, with a lower numeric value representing better visual acuity. No hypothesis testing was prespecified for this endpoint.
Time Frame: Year 2 post-implantation from second eye surgery
Population: All Implanted Analysis Set with data
Measure: Mean (Standard Deviation); unit: logMAR
Units Other Than Participants: first implanted eye
Arm/Group | Clareon IOL
Number analyzed (Participants) | 190
Number analyzed (first implanted eye) | 190
logMAR | 0.088 (0.1533)

10. Secondary Outcome: UCDVA at 2 Years Post-Implantation - Second Implanted Eye
Description: as for outcome 8
Time Frame: Year 2 post-implantation from second eye surgery
Population: All Implanted Analysis Set with data
Measure: Mean (Standard Deviation); unit: logMAR
Units Other Than Participants: second implanted eye
Arm/Group | Clareon IOL
Number analyzed (Participants) | 189
Number analyzed (second implanted eye) | 189
logMAR | 0.083 (0.1624)

11. Secondary Outcome: UCDVA at 3 Years Post-Implantation - First Implanted Eye
Description: as for outcome 9
Time Frame: Year 3 post-implantation from second eye surgery
Population: All Implanted Analysis Set
Measure: Mean (Standard Deviation); unit: logMAR
Units Other Than Participants: first implanted eye
Arm/Group | Clareon IOL
Number analyzed (Participants) | 183
Number analyzed (first implanted eye) | 183
logMAR | 0.091 (0.1614)

12. Secondary Outcome: UCDVA at 3 Years Post-Implantation - Second Implanted Eye
Description: as for outcome 8
Time Frame: Year 3 post-implantation from second eye surgery
Population: All Implanted Analysis Set with data
Measure: Mean (Standard Deviation); unit: logMAR
Units Other Than Participants: second implanted eye
Arm/Group | Clareon IOL
Number analyzed (Participants) | 182
Number analyzed (second implanted eye) | 182
logMAR | 0.086 (0.1706)

ADVERSE EVENTS:
Time Frame: Adverse events (AEs) were collected pre-treatment (Day -60 to 0) up to Day 990-1140 post-treatment/study exit. AEs were obtained through solicited and spontaneous comments from subjects and through observations by the Investigator.
Description: This analysis population includes all subjects/eyes with attempted implantation with the test article (successful or aborted after contact with the eye). "At Risk" population of pre-treatment and systemic AEs is reported in units of subjects; ocular AE population is reported in units of eyes.
Groups:
- Pretreatment: Events reported in this group occurred prior to attempted implantation with the test article
- SY60WF First Eye: Events reported in this group occurred after attempted implantation with the test article and include ocular events in the first implanted eye
- SY60WF Second Eye: Events reported in this group occurred after attempted implantation with the test article and include ocular events in the second implanted eye
- SY60WF Systemic: Events reported in this group occurred after attempted implantation with the test article
Arm/Group | Pretreatment | SY60WF First Eye | SY60WF Second Eye | SY60WF Systemic
All-Cause Mortality (participants affected / at risk) | 0/215 | 0/215 | 0/209 | 10/215
Serious Adverse Events (participants affected / at risk) | 0/215 | 6/215 | 4/209 | 31/215
Other Adverse Events (participants affected / at risk) | 0/215 | 34/215 | 39/209 | 0/215
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Pretreatment (N=215) | SY60WF First Eye (N=215) | SY60WF Second Eye (N=209) | SY60WF Systemic (N=215)
Angina pectoris (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Atrial fibrillation (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Cardiopulmonary failure (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Coronary artery disease (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Myocardial infarction (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 3 (3)
Myocardial ischaemia (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Age-related macular degeneration (Eye disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Cystoid macular oedema (Eye disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Iridocyclitis (Eye disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Macular oedema (Eye disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Retinal detachment (Eye disorders) | 0 (0) | 1 (3) | 0 (0) | 0 (0)
Retinal vein occlusion (Eye disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Rhegmatogenous retinal detachment (Eye disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Abdominal discomfort (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Diarrhoea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pancreatitis chronic (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Adverse drug reaction (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Death (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Multiple organ dysfunction syndrome (General disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Cholelithiasis (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Asymptomatic COVID-19 (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Biliary sepsis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
COVID-19 (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 3 (3)
COVID-19 pneumonia (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Influenza (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pneumonia (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pyelonephritis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Anterior capsular rupture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Fall (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hip fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Subdural haematoma (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Thermal burn (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Wrist fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Blood pressure decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Intraocular pressure increased (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hypokalaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Colon cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Lung neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Cerebellar stroke (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hydrocephalus (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Transient ischaemic attack (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Uterine prolapse (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Cholelithotomy (Surgical and medical procedures) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Intra-ocular injection (Surgical and medical procedures) | 0 (0) | 4 (7) | 2 (7) | 0 (0)
Spinal operation (Surgical and medical procedures) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Vitrectomy (Surgical and medical procedures) | 0 (0) | 1 (5) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Pretreatment (N=215) | SY60WF First Eye (N=215) | SY60WF Second Eye (N=209) | SY60WF Systemic (N=215)
Dry eye (Eye disorders) | 0 (0) | 23 (24) | 22 (22) | 0 (0)
Posterior capsule opacification (Eye disorders) | 0 (0) | 11 (11) | 19 (19) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Sponsor reserves the right of prior review of any publication or presentation of information related to the study.

DOCUMENTS (2):
  • Study Protocol (2019-11-20): https://cdn.clinicaltrials.gov/large-docs/85/NCT03316885/Prot_000.pdf
  • Statistical Analysis Plan (2019-11-21): https://cdn.clinicaltrials.gov/large-docs/85/NCT03316885/SAP_001.pdf